CLINICAL TRIAL: NCT05966896
Title: Epidural Stimulation to Restore Voluntary Movement Following Spinal Cord Injury: Spared Fibers Proof-of-concept Study
Brief Title: Epidural Stimulation to Restore Voluntary Movement Following Spinal Cord Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-0202; 1K01HD106928-01A1 (NIH)
Record Dates: First submitted 2023-07-06; First posted 2023-08-01 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Epidural stimulation with Physical Therapy (Experimental): Stimulation parameters will be optimized for each lower extremity and joint movement. During physical therapy sessions, electrode configurations may be adjusted as needed to optimize stimulation frequencies, and voltage intensity ranges to best enable voluntary control of lower extremity (ankle, knee, and hip) flexion and extension, as well as standing.
  Intensive physical therapy will consist of 3 visits per week over the course of 6 months directed by a licensed physical therapist with over a decade of experience working with individuals with spinal cord injury, and the epidural stimulator will be ON continuously during these sessions. Physical therapy will involve neurorehabilitation to facilitate voluntary lower extremity movement in the presence of stimulation, with the research participants in the supine, seated, and standing positions.
  Interventions: Device: implanted epidural stimulator

INTERVENTIONS:
Device: implanted epidural stimulator — implantable multi-programmable neurostimulation system to deliver electrical stimulation to neural targets in the spinal cord

SUMMARY:
This proof-of-concept case series will prospectively use magnetic resonance imaging (MRI) evidence of spared spinal cord neural fibers to guide the selection of 2 research participants to receive a surgically implanted epidural stimulator with the goal of restoring voluntary movement after spinal cord injury (SCI).

Because MRI evidence of spared spinal cord neural fibers demonstrated significant relationships with responsiveness to epidural stimulation in SCI in retrospective studies, the proposed study is a traditional feasibility study - a prospective investigation to be used to capture preliminary safety and effectiveness information to determine if MRI can/should be used in planning a future pivotal study.

DETAILED DESCRIPTION:
This is an investigator-initiated proof of concept study performed at the University of Colorado Anschutz Medical Campus (CU Anschutz).

This 2-case proof-of-concept study will include 2 research participants with motor-complete SCI to evaluate the performance of the Medtronic epidural stimulator for restoring voluntary movement below the level of injury.

Participants will be enrolled at CU Anschutz. Screening data will be reviewed to determine participant eligibility. Two participants who meet all inclusion criteria and none of the exclusion criteria will be entered into the study.

The following treatment regimen will be used: epidural stimulation + 6 months of intensive outpatient physical therapy.

Total duration of study participation will be 8 months.

ELIGIBILITY:
Inclusion Criteria:

1. American Spinal Injury Association Impairment Scale B spinal cord injury diagnosis
2. Beyond 6 months of injury date
3. Spinal cord injury at a level range of cervical 7 to thoracic 8 (C7-T8) with signs of upper motor neuron injury
4. 18 years or older
5. Height 5'1" to 6'3"
6. Weight 250 lbs or less
7. Sufficient upper extremity strength to manage a stability aide
8. Magnetic resonance imaging evidence of spared spinal cord neural fibers

Exclusion Criteria:

1. Claustrophobia and/or other contraindications to magnetic resonance imaging
2. Unstable or symptomatic cardiorespiratory issues, in the opinion of the investigators
3. Recent (within 3 months) history of fracture, contractures, pressure sore, deep vein thrombosis, urinary tract infection, or other infections that might interfere with interventions
4. Contraindications to epidural stimulator implantation surgery
5. Received botox injections into the lower extremities within the past 6 months
6. Pregnancy
7. Cauda Equina injury
8. Any other neurological disorder besides spinal cord injury

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
International Standards for Neurological Classification of Spinal Cord Injury lower extremity motor scores (ISNCSCI-LEMS) | at day 1, at month 7, and at month 8
  International Standards for Neurological Classification of Spinal Cord Injury lower extremity motor scores (ISNCSCI-LEMS) will be used to measure the degree of voluntary motor change. LEMS is conducted with the participant lying supine and five key muscle groups on each side are tested for their ability to contract against gravity and resistance. ISNCSCI motor testing has been shown to have adequate to excellent interrater reliability in individuals with spinal cord injury, and is a valid tool for this population.

SECONDARY OUTCOMES:
The abbreviated World Health Organization Quality of Life (WHOQOL-BREF) | at day 1, at month 7, and at month 8
  The abbreviated World Health Organization Quality of Life (WHOQOL-BREF) instrument will be used to measure the degree of participants' perception of change in quality of life after stimulator implantation. The WHOQOL-BREF assesses quality of life within the context of an individual's culture, value systems, personal goals, standards, and concerns. It has been studied and highly recommended for individuals with spinal cord injury. Scores for the abbreviated World Health Organization Quality of Life instrument range from 0 - 100, with higher scores indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew C Smith, PT, DPT, PhD, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith AC, Angeli CA, Ugiliweneza B, Weber KA 2nd, Bert RJ, Negahdar M, Mesbah S, Boakye M, Harkema SJ, Rejc E. Spinal cord imaging markers and recovery of standing with epidural stimulation in individuals with clinically motor complete spinal cord injury. Exp Brain Res. 2022 Jan;240(1):279-288. doi: 10.1007/s00221-021-06272-9. Epub 2021 Dec 2. PMID 34854934
- [Background] Rejc E, Smith AC, Weber KA 2nd, Ugiliweneza B, Bert RJ, Negahdar M, Boakye M, Harkema SJ, Angeli CA. Spinal Cord Imaging Markers and Recovery of Volitional Leg Movement With Spinal Cord Epidural Stimulation in Individuals With Clinically Motor Complete Spinal Cord Injury. Front Syst Neurosci. 2020 Oct 21;14:559313. doi: 10.3389/fnsys.2020.559313. eCollection 2020. PMID 33192348
- [Background] Harkema S, Gerasimenko Y, Hodes J, Burdick J, Angeli C, Chen Y, Ferreira C, Willhite A, Rejc E, Grossman RG, Edgerton VR. Effect of epidural stimulation of the lumbosacral spinal cord on voluntary movement, standing, and assisted stepping after motor complete paraplegia: a case study. Lancet. 2011 Jun 4;377(9781):1938-47. doi: 10.1016/S0140-6736(11)60547-3. Epub 2011 May 19. PMID 21601270
- [Background] Angeli CA, Edgerton VR, Gerasimenko YP, Harkema SJ. Altering spinal cord excitability enables voluntary movements after chronic complete paralysis in humans. Brain. 2014 May;137(Pt 5):1394-409. doi: 10.1093/brain/awu038. Epub 2014 Apr 8. PMID 24713270
- [Background] Angeli CA, Boakye M, Morton RA, Vogt J, Benton K, Chen Y, Ferreira CK, Harkema SJ. Recovery of Over-Ground Walking after Chronic Motor Complete Spinal Cord Injury. N Engl J Med. 2018 Sep 27;379(13):1244-1250. doi: 10.1056/NEJMoa1803588. Epub 2018 Sep 24. PMID 30247091